CLINICAL TRIAL: NCT03700164
Title: The Effect of Cold Exposure on the Glycaemic and Insulinaemic Responses to an Oral Glucose Load
Brief Title: The Effect of Cold Exposure on Glucose Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COGT
Record Dates: First submitted 2018-09-11; First posted 2018-10-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hyperglycemia
Keywords: Cold Exposure; Glucose Tolerance
MeSH Terms: conditions — Hyperglycemia | interventions — Temperature

STUDY DESIGN:
Intervention Model Description: It is anticipated that 32 participants will enrol in the study. Specifically, 16 participants will be healthy individuals and the other 16 will be individuals with impaired fasting glucose (5.6 mM to 6.9 mM) and/or blood glucose values 7.8-11.0 mM 2h after glucose drink consumption during the OGTT in screening. Initially, the study will investigate the effect of the cold exposure on healthy individuals, and then depending on the results in these individuals, the intervention may be tested on participants with impaired glucose metabolism.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold exposure (Experimental): Participants will be wrapped in a water-perfused suit. The temperature of the suit will be lowered to 10°C. From the onset of shivering, the participants will remain in the suit for 1 hour.
  Interventions: Other: Temperature
- Thermoneutral (Control) (Other): Participants will be wrapped in a water-perfused suit. The temperature of the suit will remain at a thermoneutral temperature (32°C) to avoid shivering and excessive sweating.
  The duration will be matched to that during the cold exposure.
  Interventions: Other: Temperature

INTERVENTIONS:
Other: Temperature — Water-perfused suit.

SUMMARY:
The purpose of the study is to evaluate the effect of cold exposure on an individual's glucose tolerance. Previous research has already shown that 10 days acclimation to a mild cold environment (14-15°C) can enhance insulin sensitivity. However, the duration in the cold environment was 6 hours per day which may not be practical for everyone. Therefore, the present study will investigate the effect of a shorter, and more intense cold exposure on an individual's glucose tolerance. It is hypothesised that cold exposure before consuming a glucose drink will enhance glucose clearance.

ELIGIBILITY:
Inclusion Criteria of healthy population:

* Signed informed consent.
* White European.
* Male.
* Age 18 - 40 years at the start of the study.
* BMI ≥ 20 and < 30 kg/m2.

Exclusion Criteria of healthy population:

* Smoking.
* Active diseases (cardiovascular, diabetes mellitus, liver, kidney, cancer or other).
* Cold-acclimated (takes daily cold baths, works in a refrigerated environment, or regular cold water swimmer).
* Unstable body weight (gain or loss > 5kg in last 3 months).
* Currently undertaking a diet.

Inclusion Criteria of prediabetes population:

* Signed informed consent.
* White European.
* Male or female.
* Women should be postmenopausal or use hormonal contraceptives.
* Age 30 - 75 years at the start of the study.
* BMI ≥ 25 and < 35 kg/m2.
* Generally healthy, no medication use that interferes with metabolism. If volunteers need medication (e.g. statin drugs, NSAIDs), it will be reviewed with the dependent physician on an individual basis.
* Impaired fasting glucose (5.6 mM to 6.9 mM) and/or blood glucose values 7.8-11.0 mM 2h after glucose drink consumption during OGTT in screening.

Exclusion Criteria of prediabetes population:

* Smoking.
* Active diseases (cardiovascular, diabetes mellitus, liver, kidney, cancer or other).
* Cold-acclimated (takes daily cold baths, works in a refrigerated environment, or regular cold water swimmer).
* Unstable body weight (gain or loss > 5kg in last 3 months).
* Currently undertaking a diet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Glucose and insulin concentrations in response to an oral glucose load | 3 hours post glucose drink, measured 90 minutes after the cold exposure

SECONDARY OUTCOMES:
Energy expenditure measured using indirect calorimetry | 30 minutes before and during the 1 hour of cold exposure
Core temperature measured using a telemetric pill | 30 minutes before and during the 1 hour of cold exposure
Skin blood flow measured using laser doppler flowmetry | 30 minutes before and during the 1 hour of cold exposure
Shivering activity assessed using surface electromyography | 30 minutes before and during the 1 hour of cold exposure
Systolic and diastolic blood pressure measured using an automatic blood pressure device | 30 minutes before and during the 1 hour of cold exposure
Thermal sensation | 30 minutes before and during the 1 hour of cold exposure
  How warm or cold the participant perceives the environment. Assessed with a visual analogue scale (scale ranging from cold to hot).
Skin temperature measured using iButtons | 30 minutes before and during the 1 hour of cold exposure
Heart rate measured using chest heart rate monitor sensor | 30 minutes before and during the 1 hour of cold exposure
Comfort | 30 minutes before and during the 1 hour of cold exposure
  How comfortable or uncomfortable the participant perceives the environment. Comfort assessed with a visual analogue scale (scale ranging from very comfortable to very uncomfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Wouter van Marken Lichtenbelt, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands